CLINICAL TRIAL: NCT01966705
Title: Self-help Based Cognitive Behavior Therapy for Health Anxiety Delivered Via the Internet or in Book Form - the Effect of Administration Strategy and Therapist Contact: a Randomized Controlled Trial
Brief Title: Cognitive Behavior Therapy for Health Anxiety: A Comparison of Three Forms of Self-help
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Hedman, phd, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: InterBib
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Severe Health Anxiety; Somatic Symptom Disorder; Illness Anxiety Disorder
Keywords: severe health anxiety; somatic symptom disorder; illness anxiety disorder; cognitive behavior therapy; bibliotherapy; internet; exposure
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Therapist-guided Internet-based Cognitive Behavior Therapy (Experimental): Cognitive Behavior Therapy delivered via the Internet: 12 weeks, supported self-help
  Interventions: Behavioral: Cognitive Behavior Therapy, exposure and response prevention (Internet, guided)
- Unguided Internet-based Cognitive Behavior Therapy (Experimental): Cognitive Behavior Therapy delivered via the Internet: 12 weeks, self-help only
  Interventions: Behavioral: Cognitive Behavior Therapy, exposure and response prevention (Internet, unguided)
- Cognitive Behavior Therapy-based bibliotherapy (Experimental): Cognitive Behavior Therapy delivered in book form: 12 weeks, self-help only
  Interventions: Behavioral: Cognitive Behavior Therapy, exposure and response prevention (Book, unguided)
- Waiting-list condition (No Intervention): No intervention: 12 weeks

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy, exposure and response prevention (Internet, guided) — This intervention entails different exercises aimed at exposure to health anxiety stimuli.
  Participants are guided by a therapist. Treatment is delivered via the Internet.
  Arms: Therapist-guided Internet-based Cognitive Behavior Therapy
Behavioral: Cognitive Behavior Therapy, exposure and response prevention (Internet, unguided) — This intervention entails different exercises aimed at exposure to health anxiety stimuli.
  Participants are not guided by a therapist. Treatment is delivered via the Internet.
  Arms: Unguided Internet-based Cognitive Behavior Therapy
Behavioral: Cognitive Behavior Therapy, exposure and response prevention (Book, unguided) — This intervention entails different exercises aimed at exposure to health anxiety stimuli.
  Participants are not guided by a therapist. Treatment is delivered in book form.
  Arms: Cognitive Behavior Therapy-based bibliotherapy

SUMMARY:
Background

Severe health anxiety, Somatic symptom disorder or Illness anxiety disorder according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5), is associated with considerable personal distress, functional disability and societal costs. Several studies have demonstrated the efficacy of Cognitive Behavior Therapy (CBT) for severe health anxiety, both on anxiety itself and on secondary symptom measures (for example of depression). One published randomized controlled trial (RCT) has examined the feasibility of delivering CBT for severe health anxiety via the Internet as a form of guided self help. Participants had contact with a therapist via an e-mail-like system throughout the treatment. This approach yielded results superior to a waiting-list condition, thus potentially greatly increasing the availability of psychological treatment. However, more studies on the effects of Internet-delivered CBT are warranted (NCT01673035 being one). Additionally, little is known about the active ingredients and mechanisms of change involved in Internet-delivered CBT. For example, the significance of therapist support in relation to treatment outcomes remains to be determined. CBT-based self-help literature, so called bibliotherapy, has shown great promise in the treatment of several anxiety disorders, including panic disorder and social anxiety disorder. Two small pilot studies have indicated that bibliotherapy with no or minimal therapist contact could be suitable for treating health anxiety.

Aim of the study

The aim of the present RCT is to compare therapist-guided Internet-delivered CBT (n=33), Internet-delivered CBT without therapist guidance (n=33), CBT-based bibliotherapy without therapist guidance (n=33) and a waiting-list control condition (n=33) for adult participants with severe health anxiety.

Participants in all treatment programs are expected to be significantly improved on measures of health anxiety, compared to participants allocated to the waiting-list condition.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of severe health anxiety (somatic symptom disorder or illness anxiety disorder) according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5)
* At least 18 years old
* Able to read and write in Swedish

Exclusion Criteria:

* Other primary axis-I disorder
* Ongoing substance abuse or addiction
* Current or previous episode of psychosis or bipolar disorder
* Severe major depressive disorder
* Higher than 5 on the suicidality scale of the Mini International diagnostic Interview
* Non-stable antidepressant medication (changed during the last 2 months) or not agreeing to keep dosage constant throughout the study
* Ongoing concurrent psychological treatment for severe health anxiety
* Having received previous high quality Cognitive Therapy or Cognitive Behavior Therapy during the recent year
* Ongoing serious somatic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Health Anxiety Inventory (HAI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in HAI at post-treatment and follow-ups compared to baseline

SECONDARY OUTCOMES:
Illness Attitude Scale (IAS) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in IAS at post-treatment and follow-ups compared to baseline
Whiteley Index (WI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in WI at post-treatment and follow-ups compared to baseline
Montgomery-Åsberg Depression Rating Scale - Self report (MADRS-S) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in MADRS-S at post-treatment and follow-ups compared to baseline
Beck Anxiety Inventory (BAI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in BAI at post-treatment and follow-ups compared to baseline
Anxiety Sensitivity Index (ASI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in ASI at post-treatment and follow-ups compared to baseline
Sheehan Disability Scale (SDS) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in SDS at post-treatment and follow-ups compared to baseline
Trimbos and institute of medical technology assessment cost questionnaire (TIC-P) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in TIC-P at post-treatment and follow-ups compared to baseline
Euroqol-5D (EQ-5D) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in EQ-5D at post-treatment and follow-ups compared to baseline
Obsessive Compulsive Inventory Revised (OCI-R) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Only for assessing the sample on this symptom domain
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Only for assessing the sample on this symptom domain
Alcohol Use Disorders Identification Test (AUDIT) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in AUDIT at post-treatment and follow-ups compared to baseline
Insomnia Severity Index (ISI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in ISI at post-treatment and follow-ups compared to baseline
Self-rated health 5 (SRH-5) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in SRH-5 at post-treatment and follow-ups compared to baseline
The Swedish Scales of Personalities | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in The Swedish Scales of Personalities at post-treatment and follow-ups compared to baseline
Quality of Life Inventory (QOLI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in QOLI at post-treatment and follow-ups compared to baseline

OTHER OUTCOMES:
Psychological mediators | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Assessment of whether these mediators will precede change in outcome during the treatment. Mediators will be assessed using sub scales of the Health Anxiety Inventory, and the Insomnia Severity Index, Perceived Competence Scale, Working Alliance Inventory, Five Facet Mindfulness Questionnaire, Acceptance and Flexibility, and Somatosensory Amplification Scale
The treatment credibility scale | Weeks 2 and 8
  For assessing treatment credibility and expectancy of improvement

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hedman, phd, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Background] Hedman E, Andersson E, Lindefors N, Andersson G, Ruck C, Ljotsson B. Cost-effectiveness and long-term effectiveness of internet-based cognitive behaviour therapy for severe health anxiety. Psychol Med. 2013 Feb;43(2):363-74. doi: 10.1017/S0033291712001079. Epub 2012 May 21. PMID 22608115
- [Background] Jones FA. The role of bibliotherapy in health anxiety: an experimental study. Br J Community Nurs. 2002 Oct;7(10):498-504. doi: 10.12968/bjcn.2002.7.10.10662. PMID 12399701
- [Background] Buwalda FM, Bouman TK. Cognitive-behavioural bibliotherapy for hypochondriasis: a pilot study. Behav Cogn Psychother. 2009 May;37(3):335-40. doi: 10.1017/S1352465809005293. Epub 2009 May 6. PMID 19416560
- [Background] Salkovskis PM, Rimes KA, Warwick HM, Clark DM. The Health Anxiety Inventory: development and validation of scales for the measurement of health anxiety and hypochondriasis. Psychol Med. 2002 Jul;32(5):843-53. doi: 10.1017/s0033291702005822. PMID 12171378
- [Background] Furer P, Walker JR. Treatment of Hypochondriasis with Exposure. Journal of Contemporary Psychotherapy 35(3): 251-267, 2005.
- [Derived] Axelsson E, Osterman S, Hedman-Lagerlof E. Joint factor analysis and approximate equipercentile linking of common trait health anxiety measures: a cross-sectional study of the 14-, 18- and 64-item health anxiety inventory, the illness attitude scale, and the 14-item Whiteley Index. BMC Psychiatry. 2023 Sep 6;23(1):658. doi: 10.1186/s12888-023-05151-7. PMID 37674135
- [Derived] Hedman-Lagerlof E, Axelsson E, Andersson E, Ljotsson B, Andreasson A, Lekander M. The impact of exposure-based cognitive behavior therapy for severe health anxiety on self-rated health: Results from a randomized trial. J Psychosom Res. 2017 Dec;103:9-14. doi: 10.1016/j.jpsychores.2017.09.013. Epub 2017 Sep 28. PMID 29167052
- [Derived] Hedman E, Axelsson E, Andersson E, Lekander M, Ljotsson B. Exposure-based cognitive-behavioural therapy via the internet and as bibliotherapy for somatic symptom disorder and illness anxiety disorder: randomised controlled trial. Br J Psychiatry. 2016 Nov;209(5):407-413. doi: 10.1192/bjp.bp.116.181396. Epub 2016 Aug 4. PMID 27491531